CLINICAL TRIAL: NCT03937726
Title: Boiled Peanut Immunotherapy for the Treatment of Peanut Allergy: A Non-inferiority Study
Brief Title: Boiled Peanut Immunotherapy for the Treatment of Peanut Allergy
Acronym: BOPI-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19SM5033
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: IgE Mediated Peanut Allergy; Peanut Hypersensitivity
Keywords: Peanut allergy; Desensitisation; Safety
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Masking Description: Primary outcome will be assessed by double-blind, placebo-controlled food challenge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boiled peanut Oral Immunotherapy (Experimental): Desensitisation using boiled peanut
  Interventions: Other: Boiled peanut
- Conventional Oral immunotherapy (Active Comparator): Desensitisation using defatted peanut flour
  Interventions: Other: Defatted roasted peanut flour

INTERVENTIONS:
Other: Boiled peanut — Desensitisation using boiled peanut for induction and initial updosing
  Arms: Boiled peanut Oral Immunotherapy
Other: Defatted roasted peanut flour — Desensitisation using defatted peanut flour for induction and initial updosing
  Arms: Conventional Oral immunotherapy

SUMMARY:
Peanut allergy is the most common cause of severe allergic reactions to food. Onset is common in childhood, but in contrast to other food allergies such as cow's milk and egg, peanut allergy tends to persist into adulthood. It is associated with a significant impact on quality of life, both for the affected individual and their family.

There is no current cure for peanut allergy. Oral peanut immunotherapy (OIT) using defatted, roasted peanut flour has been demonstrated to offer potential in this regard, but is associated with significant and frequent reactions and can cause life-threatening allergic symptoms.

The investigators have previously demonstrated that the processing of peanuts through boiling results in a relatively hypoallergenic product due to the loss of key allergenic components from peanut into the water. This has been tested in a recently-completed Phase 2b/3 trial (The BOPI Study, Clinicaltrials.gov NCT02149719; HRA reference 15/LO/0287): 47 children/ young people with peanut allergy confirmed at double-blind, placebo-controlled food challenge (DBPCFC) were randomised (2:1) to receive either oral immunotherapy (updosing using boiled peanut for ~6 months, followed by maintenance with roasted peanut) or standard treatment (allergen avoidance). Participants underwent repeat DBPCFC at 12 months to assess response, following which peanut OIT was stopped and sustained unresponsiveness assessed after 4 weeks (4SU). 24/32 participants (100% per protocol) achieved the primary outcome of desensitisation to >1.44g peanut protein (approximately 6-8 peanuts, p<0.0001); of those 14 tolerated >4.4g peanut protein. 13/24 participants achieved 4SU. There was no significant change in threshold in the control group (p>0.05). Boiled peanut OIT had a favourable safety profile, with under 2% of doses associated with gastrointestinal symptoms.

The BOPI-2 study is a non-inferiority study to demonstrate that boiled peanut is at least as effective as peanut flour in treating children with peanut allergy. The study will compare the rate of adverse events and other safety outcomes between these two interventions, and assess the immunological mechanisms involved, a secondary aim being to develop clinically-useful predictors for identifying individuals likely to undergo successful desensitisation.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-18 years (enrolment up to a participant's 19th birthday).
* Past history consistent with IgE-mediated peanut allergy
* Allergic to ≤1.44 g peanut protein (approx. 6 peanuts) at baseline double-blind placebo-controlled food challenge, prior to treatment allocation
* Tolerates at least 1/8 boiled peanut (boiled for 4 hours) at open food challenge at screening.
* Written informed consent of parent/legal guardian and patient assent.

Exclusion Criteria:

* Required previous admission to an intensive care unit for management of an allergic reaction to peanut.
* Clinically significant chronic illness (other than asthma, rhinitis or eczema).
* Undergoing subcutaneous or sublingual immunotherapy to respiratory allergens, and not yet established on maintenance dosing for at least 3 months.
* Undergoing oral immunotherapy for food allergy and within the first year of treatment.
* Subjects receiving anti-IgE therapy, oral immunosuppressants, beta-blocker or ACE inhibitor.
* Tolerance to ≥1.44 g peanut protein (approx. 6 peanuts) at initial DBPCFC during screening.
* Dose-limiting symptoms to 1/8 boiled peanut (boiled for 4 hours) at screening.
* Poorly controlled asthma within the previous 3 months (as defined by clinician judgement with reference to the ICON consensus ), or asthma requiring treatment with >5 days oral corticosteroids within the previous 3 months.
* Pregnancy
* Unwilling or unable to fulfil study requirements

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Desensitisation to >1.4g (roasted) peanut protein at food challenge | 12 months
  The proportion of participants who tolerate 1.44g (or more) roasted peanut protein (equivalent to ≥ 6 roasted peanuts) after 12 months of OIT, as assessed by DBPCFC, in each treatment group.

SECONDARY OUTCOMES:
Adverse events | 12 months
  The proportion of participants experiencing adverse events classified as mild non-transient symptoms or more severe during updosing and maintenance in each treatment group.
Other safety outcomes | 12 months
  Rates of adverse events by type / organ involved in each treatment group
Change in Health-related quality of life (HRQL) from baseline - assessed using FAQLQ | 6,12 and 13+ months
  Change in HRQL measures at 6, 12 and 13 months from baseline, as assessed in study participants and their parent/carer using the following validated questionnaire:
  - Food Allergy Quality of Life Questionnaire (FAQLQ) (reference Muraro et al, 2014)
Change in Health-related quality of life (HRQL) from baseline - assessed using FAIM | 6,12 and 13+ months
  Change in HRQL measures at 6, 12 and 13 months from baseline, as assessed in study participants and their parent/carer using the following validated questionnaire:
  - Food Allergy Independent Measure (FAIM) (see Muraro et al, 2014)
Change in Health-related quality of life (HRQL) from baseline - assessed using standardized instrument (EQ-5D) | 6,12 and 13+ months
  Change in HRQL measures at 6, 12 and 13 months from baseline, as assessed using the following validated questionnaire:
  - EQ-5D - a standardized instrument for use as a measure of health outcome. (Further details at https://euroqol.org/)
Change in Health-related quality of life (HRQL) from baseline - assessed using standardized instrument (CHU-9D) | 6,12 and 13+ months
  Change in HRQL measures at 6, 12 and 13 months from baseline, as assessed using the following validated questionnaire:
  - CHU-9D (The Child Health Utility 9D) - also a standardized instrument for use as a measure of health outcome. (Further details at https://www.sheffield.ac.uk/scharr/sections/heds/mvh/paediatric)
Change in self-efficacy after each phase of immunotherapy | 6,12 and 13+ months
  Change in self-efficacy at 6, 12 and 13 months from baseline, as assessed in study participants and their parent/carer using validated questionnaire.
Immunological outcome: skin prick test | 12 months
  Change in skin prick test wheal (mm) and end-point titration skin prick test between baseline and post immunotherapy
Immunological outcome: Allergen-specific IgE | 12 months
  Change in allergen-specific IgE (kUa/l) between baseline and post immunotherapy

OTHER OUTCOMES:
Sustained unresponsiveness after 4 weeks cessation of maintenance OIT | After 1 year of OIT
  Rate of sustained unresponsiveness after 4 weeks cessation of maintenance OIT at 1 year.
Sustained unresponsiveness after 12+ weeks cessation of maintenance OIT | After 1 year of OIT
  Rate of sustained unresponsiveness after 12+ weeks cessation of maintenance OIT at 1 year, in those participants who demonstrate sustained unresponsiveness at 4 weeks off maintenance OIT.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, FRACP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust (St. Mary's Hospital), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muraro A, Dubois AE, DunnGalvin A, Hourihane JO, de Jong NW, Meyer R, Panesar SS, Roberts G, Salvilla S, Sheikh A, Worth A, Flokstra-de Blok BM; European Academy of Allergy and Clinical Immunology. EAACI Food Allergy and Anaphylaxis Guidelines. Food allergy health-related quality of life measures. Allergy. 2014 Jul;69(7):845-53. doi: 10.1111/all.12405. Epub 2014 May 2. PMID 24785644
- See also: Related Info — https://www.imperial.ac.uk/news/190335/promising-peanut-trial-offers-hope-children/